CLINICAL TRIAL: NCT06272903
Title: The Immediate Effect of Benzocaine 20% Topical Anesthesia on Pain Levels When Placing Elastomeric Orthodontic Separators in Children Receiving Hall Technique Crowns: A Randomized Control Trial
Brief Title: Effect of Benzocaine 20% Topical Anesthesia on Pain Levels When Placing Separators in Children Receiving Hall Technique Crowns
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Simran Kaur Sura, Resident - Pediatric Dentistry, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBRU IRB-2023-228
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-02

CONDITIONS: Effect of Benzocaine on Pain
MeSH Terms: interventions — Benzocaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benzocaine 20% Topical Anesthesia Arm (Experimental): Participants will be assigned this arm either to their right or left hand side of their mouth. They will receive benzocaine 20% topical anesthesia prior to the placement of elastomeric orthodontic separators.
  The topical anesthesia will be applied according to standard clinical practice. Pain and discomfort levels associated with the placement of separators will be assessed immediately after the procedure.
  Interventions: Drug: 20% benzocaine, topical anesthetic
- Placebo (Children's Toothpaste) Arm (Placebo Comparator): The other side of the mouth will receive a placebo, which consists of children's toothpaste, prior to the placement of elastomeric orthodontic separators.
  The toothpaste will be applied according to standard clinical practice. Pain and discomfort levels associated with the placement of separators will be assessed immediately after the procedure.
  Interventions: Other: Children's Toothpaste

INTERVENTIONS:
Drug: 20% benzocaine, topical anesthetic — Indicated as a topical anesthetic for use on oral mucosa prior to local anesthetic injections, scaling and prophylaxis. Also useful to relieve discomfort associated with taking impressions and intra- oral radiographs.
  The benzocaine topical anesthetic will be applied according to standard clinical practice, aiming to provide local anesthesia to the treatment site and minimize discomfort during the procedure (placing elastomeric orthodontic separators).
  Arms: Benzocaine 20% Topical Anesthesia Arm
Other: Children's Toothpaste — Strawberry-flavored children's toothpaste available in Dubai, UAE.
  Arms: Placebo (Children's Toothpaste) Arm

SUMMARY:
The goal of this RCT is to investigate the immediate effect of benzocaine 20% topical anesthesia on initial pain and discomfort levels associated with the placement of elastomeric orthodontic separators in children who are receiving Hall Technique crowns on primary molars, among children who have attended the Pediatric Dentistry Department, Dubai Dental Hospital (DDH), Mohammed Bin Rashid University (MBRU) in Dubai, the United Arab Emirates (UAE).

DETAILED DESCRIPTION:
The primary objective of this RCT is to assess the immediate effect of benzocaine 20% topical anesthesia on the initial pain and discomfort experienced during the placement of elastomeric orthodontic separators in pediatric patients undergoing Hall Technique crowns for their primary molars. This study will be conducted among children aged 4-10 years old, receiving dental care at the Pediatric Dentistry Department of Dubai Dental Hospital (DDH), Mohammed Bin Rashid University (MBRU) in Dubai, United Arab Emirates (UAE).

The research will involve recruiting a sample of 32 pediatric patients aged between 4 and 10 years who require 2 Hall Technique crowns on their primary molars and are scheduled to undergo the placement of elastomeric orthodontic separators as part of their treatment. The participants will be randomly assigned to receive benzocaine 20% topical anesthesia prior to separator placement on either the right or left side of their mouth, and the other side receiving a placebo (e.g., children's toothpaste) before separator placement.

Data collection: following the placement of elastomeric orthodontic separators, participants will be asked to rate their pain and discomfort levels immediately after the procedure using the Wong-Baker FACES Pain Rating Scale.

In addition to pain and discomfort assessments, demographic data (e.g., age, gender) and clinical information (e.g., specific teeth undergoing treatment) will be collected for each participant. The study will employ rigorous blinding procedures to ensure that the participants are unaware of the assigned treatment (benzocaine or placebo) during the procedure and data collection phases. The principle investigator will only be aware of which side of the mouth will be receiving benzocaine just before the procedure via a sealed envelope randomisation.

Statistical analyses will be conducted to compare the pain and discomfort levels between the two treatment groups. The findings of this study will contribute valuable insights into the efficacy of benzocaine 20% topical anesthesia in managing pain associated with elastomeric orthodontic separator placement in pediatric dental patients undergoing Hall Technique crown procedures. Ultimately, the results will inform clinical practice and improve the quality of care provided to pediatric patients undergoing dental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children with asymptomatic non pulpally involved carious primary molars who meet the indications of the HT in Dubai Dental Hospital.
* Children who require same tooth bilateral HT Crowns in either bilateral or diagonal pattern.
* Healthy male and female children, aged 4-10 years (ASA 1) with no conditions that affect sensory input/reaction.
* Children who are verbal and able to communicate.
* Not taking any painkillers, or other drugs that would influence with their pain perception.
* Cooperative children.
* Parents or guardians who consent for their children to be enrolled in the trial.

Exclusion Criteria:

* Children who are indicated for bilateral HT but do not require EOS, due to pre-existing interdental spaces.
* Children who are indicated for bilateral HT but parents prefer or indicate preference for the Modified HT.
* Children with allergies to nickel or other metal components that constitute a PMC.
* Those with reported allergies to topical or local anesthetic.
* Children with special health care needs or those who are non-verbal and are unable to communicate their pain levels.
* Children/parents/guardians not willing to participate in the study.
* Patients that require treatment under conscious sedation or general anesthesia.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Immediate Pain Levels | Immediate (within 30 seconds of placing elastomeric orthodontic separators)
  The primary outcome measure is the immediate pain and discomfort experienced by children following the placement of EOSs in the context of placing them before the Hall Technique Crown is placed. It will be assessed using a standardized pain scale (Wong-Baker Faces pain scale) where the participants will rate their pain levels immediately after the procedure.

SECONDARY OUTCOMES:
Patient Satisfaction During Procedure | Immediate (within 30 seconds)
  I will be gathering feedback from the children regarding their overall satisfaction with the procedure by using the Wong-Baker Faces pain scale. This will enable us to gauge the acceptability of placing the elastomeric orthodontic separators.

CONTACTS AND LOCATIONS:
Overall Officials: Simran Kaur Sura, Principal Investigator — Mohammed Bin Rashid University of Medicine and Health Sciences
Locations (1):
- Mohammed Bin Rashid University Of Medicine and Health Sciences, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussein I, Al Halabi M, Kowash M, Salami A, Ouatik N, Yang YM, Duggal M, Chandwani N, Nazzal H, Albadri S, Roberts A, Al-Jundi S, Nzomiwu C, El Shahawy O, Attaie A, Mohammed O, Al-Sane M. Use of the Hall technique by specialist paediatric dentists: a global perspective. Br Dent J. 2020 Jan;228(1):33-38. doi: 10.1038/s41415-019-1100-2. PMID 31925371
- [Background] Boyd DH, Foster Page LA, Moffat SM, Thomson WM. Time to complain about pain: Children's self-reported procedural pain in a randomised control trial of Hall and conventional stainless steel crown techniques. Int J Paediatr Dent. 2023 Jul;33(4):382-393. doi: 10.1111/ipd.13059. Epub 2023 Mar 16. PMID 36841968
- [Background] Lee HS. Recent advances in topical anesthesia. J Dent Anesth Pain Med. 2016 Dec;16(4):237-244. doi: 10.17245/jdapm.2016.16.4.237. Epub 2016 Dec 31. PMID 28879311
- [Background] Aghababaie ST, Monteiro J, Stratigaki E, Ashley PF. Techniques for effective local anaesthetic administration for the paediatric patient. Br Dent J. 2020 Dec;229(12):779-785. doi: 10.1038/s41415-020-2453-2. Epub 2020 Dec 18. PMID 33339924
- [Background] Bird SE, Williams K, Kula K. Preoperative acetaminophen vs ibuprofen for control of pain after orthodontic separator placement. Am J Orthod Dentofacial Orthop. 2007 Oct;132(4):504-10. doi: 10.1016/j.ajodo.2006.11.019. PMID 17920504
- [Background] Farzan A, Khaleghi K. The Effectiveness of Low-Level Laser Therapy in Pain Induced by Orthodontic Separator Placement: A Systematic Review. J Lasers Med Sci. 2021 Jun 24;12:e29. doi: 10.34172/jlms.2021.29. eCollection 2021. PMID 34733752
- [Background] Al-Melh MA, Nada A, Badr H, Andersson L. Effect of an Anesthetic Chewing Gum on the Initial Pain or Discomfort from Orthodontic Elastomeric Separator Placement. J Contemp Dent Pract. 2019 Nov 1;20(11):1286-1292. PMID 31892680
- [Background] Eslamian L, Borzabadi-Farahani A, Edini HZ, Badiee MR, Lynch E, Mortazavi A. The analgesic effect of benzocaine mucoadhesive patches on orthodontic pain caused by elastomeric separators, a preliminary study. Acta Odontol Scand. 2013 Sep;71(5):1168-73. doi: 10.3109/00016357.2012.757358. Epub 2013 Jan 10. PMID 23301559
- [Background] Meechan JG. Intraoral topical anesthesia. Periodontol 2000. 2008;46:56-79. doi: 10.1111/j.1600-0757.2008.00231.x. No abstract available. PMID 18201346
- [Background] Falci SG, Marques LS. CONSORT: when and how to use it. Dental Press J Orthod. 2015 May-Jun;20(3):13-5. doi: 10.1590/2176-9451.20.3.013-015.ebo. No abstract available. PMID 26154451
- [Background] Garrocho-Rangel A, Ruiz-Rodriguez S, Gaitan-Fonseca C, Pozos-Guillen A. Randomized Clinical Trials in Pediatric Dentistry: Application of Evidence-Based Dentistry through the CONSORT Statement. J Clin Pediatr Dent. 2019;43(4):219-230. doi: 10.17796/1053-4625-43.4.1. Epub 2019 May 16. PMID 31094627
- [Background] Eslamian L, Kianipour A, Mortazavi SAR. The Analgesic Efficacy of 5% Naproxen Gel for Pain Associated with Orthodontic Separator Placement: A Randomized Double-Blind Controlled Trial. Anesth Pain Med. 2017 Mar 8;7(2):e42708. doi: 10.5812/aapm.42708. eCollection 2017 Apr. PMID 28824857
- Available data/document: Study Protocol: MBRU IRB-2023-228 — http://www.mbru.ac.ae